CLINICAL TRIAL: NCT01974414
Title: Cedar Honey in Treatment of Oral Lichen Planus: a Randomized Clinical Trial
Brief Title: Cedar Honey in Oral Lichen Planus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pegah Mosannen Mozafari, Assistant professor of Oral medicine, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 900166
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Erosive and Atrophic Oral Lichen Planus
Keywords: oral lichen planus; cedar honey; atrophic; erosive; pain; treatment; clinical trial
MeSH Terms: conditions — Lichen Planus, Oral; Atrophy; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cedar honey (Active Comparator): The two study groups were provided with standard treatment(dexamethasone and Fluconazole).The Case group(A) received cedar honey, 20 ml 3 times daily by swish and swallow technique, in addition to the standard treatment .
  Interventions: Drug: orally administered cedar honey
- control group (No Intervention): the control group (B) only received standard treatment(Dexametazone and Fluconazole).

INTERVENTIONS:
Drug: orally administered cedar honey
  Arms: cedar honey

SUMMARY:
The study aimed to evaluate the effect of cedar honey in treatment of erosive and atrophic oral lichen planus ( a common oral problem).

ELIGIBILITY:
Inclusion Criteria:

1. clinically and histopathologically confirmed oral lichen planus without dysplasia in histopathologic evaluation
2. Severity of pain≥2 (VAS score)
3. Severity of lesions≥2 (tong prasom criteria)
4. absence of any treatment in the last month
5. absence of kidney or liver diseases( due to systemic administration of fluconazole to both groups)

Exclusion Criteria:

1. evidence of lichenoid reaction in clinical or histopathologic assessment
2. loss of follow up
3. pregnant patients
4. diabetic patients
5. any other mucosal disease
6. any severe systemic disease
7. patients who refuse doctor's advice
8. any unexpected adverse effect of honey

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
severity of lesions | 4 weeks
  severity of lesions due to thong prasom criteria

SECONDARY OUTCOMES:
size of lesions | 4 weeks
  A sterile caulis was used to measure the maximum diameter of erosive and atrophic lesions and the maximum width perpendicular to the maximum diameter was recorded.

OTHER OUTCOMES:
pain of lesions | 4 weeks
  Pain or burning sensation was assessed by using a visual analog scale (VAS). Patients marked the point from 0(no pain) to 10(extreme pain) representing their present pain perception

CONTACTS AND LOCATIONS:
Overall Officials: Majid Sanatkhani, Assistant Professor, Study Director — Mashhad University of Medical Sciences
Locations (1):
- Oral Medicine Department of Mashhad dental School,Oral and Maxillofacial diseases research center, Mashhad, Khorasan Razavi, Iran